CLINICAL TRIAL: NCT00735657
Title: Anesthesia for PPV Using Insulin Needle
Brief Title: Anesthesia for Pars Plana Vitrectomy (PPV) With Insulin Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rp0822
Record Dates: First submitted 2008-07-01; First posted 2008-08-15 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Retinal Disorders
Keywords: Efficiency; Pars; Plana; Vitrectomy
MeSH Terms: conditions — Retinal Diseases | interventions — Needles

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Control
  Interventions: Device: needle; Procedure: Pars Plana Vitrectomy
- Group 2 (Active Comparator): Block with short needle
  Interventions: Device: needle; Procedure: Pars Plana Vitrectomy

INTERVENTIONS:
Device: needle — Peribulbar blockade with standard (25 mm) needle
  Other Names: Peribulbar blockade with standard needle
  Arms: Group 1
Device: needle — Peribulbar blockade with short (12.5 mm) needle
  Other Names: Peribulbar blockade with short needle
  Arms: Group 2
Procedure: Pars Plana Vitrectomy — Peribulbar block
  Other Names: Extraconal block

SUMMARY:
Periocular blockade with 12.5 mm needle is as effective as block with 25 mm needle for patients undergoing Pars Plana Vitrectomy.

DETAILED DESCRIPTION:
The author wants to see the effect of short needle in patients undergoing retinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing pars plana vitrectomy under local anesthesia

Exclusion Criteria:

* Patients allergic to local anesthetic solutions
* With local sepsis
* Serious impairment of coagulation
* Orbital abnormalities
* Unable to cooperate in maintaining a relatively motionless supine position
* Who refused the anesthetic technique

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of insulin needle. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD, Principal Investigator — KKESH
Locations (1):
- King Khaled Eye Specialist hospital, Riyadh, Saudi Arabia